



## Menoufia University Faculty Of Medicine Research Ethics Committee

## **Institutional Review Board**

Assessment of a study protocol

Department: Anesthesiology, Intensive care and pain management

**Title:** Analgesic Efficacy of Combined Lumbar Erector Spinae Plane Block and Pericapsular Nerve Group Block in Patients Undergoing Hip Surgeries

| | | | *************************************** | |
|---|---|---|---|---|
| - | Approved | | | |
| - | Need changes | | | |
| Aim<br>comb | of the study:<br>ined LESPB and | evaluation of the postoperative analgesic of PENG block after hip surgeries. | efficacy of | |
| - | Approved Need changes | | | |
| Resea | arch Methodolo | gy and sample size calculations: (36 cases). | | |
| - | Approved Need changes | | | |
| Statistical Methods: | | | | |
| - | Approved Need changes | | | |
| Decis | ion: | | <u> </u> | _ |
| - Ap | Approved after Disapproved | IRB approved number and date 2/2023 amendment Signature | ANET 6 | 2 |
| | | 8 | 1 | |